CLINICAL TRIAL: NCT04683302
Title: 3D Biplane vs Conventional 2D Ultrasound Guided Internal Jugular VEin caNnulation in CardiotHoracic surgerY Patients
Brief Title: 3D Guided Internal Jugular Vein Catheterization
Acronym: 3D Givenchy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, Harm Scholten, MD, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3DJUG
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Catheter Related Complication; Ultrasound; Complications
Keywords: ultrasound; internal jugular vein; cardiothoracic surgery

STUDY DESIGN:
Intervention Model Description: randomized clinical trial (RCT)
Who Masked: Participant, Outcomes Assessor
Masking Description: coded (e)crf's and anonymized and coded ultrasound clips
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- control (Active Comparator): conventional 2D guided internal jugular vein catheterization
  Interventions: Device: 2D US catheterization
- intervention (Experimental): 3D biplanar guided internal jugular vein catheterization
  Interventions: Device: 3DUS biplanar catheterization

INTERVENTIONS:
Device: 3DUS biplanar catheterization — biplanar view of both short and long axis view of the internal jugular vein improves anatomical awareness and potentially improves safety of venous catheterization
  Arms: intervention
Device: 2D US catheterization — 2D short axis internal jugular vein catheterization
  Arms: control

SUMMARY:
Central venous catheterization through the jugular vein is a standard procedure for cardiothoracic surgical patients. Ultrasound (US) guidance is preferred and compared to traditional landmark approach decreases complications and increases success rate. Both long and short axis views are used for obtaining access, both with their own advantages and shortcomings. Complications have also not completely diminished with the use of US. The investigators propose a new technique using 3D biplanar imaging, combining advantages from both long and short axis views in one image, enabling more successful procedures and a lower complication rate

DETAILED DESCRIPTION:
Central venous catheters (CVC) are frequently placed in patients who are scheduled for cardiothoracic surgery (ICU). Ultrasound (US) guidance has consistently shown to not only improve success rate of procedures, but also to decrease complications with most benefit for the jugular vein. However, serious adverse events still occur despite US guidance Conventional two dimensional ultrasound (2D US) guided access if performed in either the short axis or long axis view, with both approaches having their own limitations. Using short axis view, the operator is never certain of the position of the needle tip as the shaft of the needle is not distinguishable from the tip in this view. Structures not (yet) visible in the US screen can already be punctured, or a vessel can be entered at a different position than preferred. A possible mechanism through which carotid artery puncture can happen is the posterior wall puncture4.

For long axis view, with proper technique the needle is viewed entirely during the procedure. However, this requires extensive experience and the overview of surrounding structures is lost.Multiple attempts at improving US guided venous access have been tried, such as oblique visualization or alternating short and long axis views but those approaches still have their shortcomings.

Three dimensional ultrasound (3D US) has a theoretical advantage of increased anatomical awareness, but evidence of improvement in needle based procedures is scarce.

Recently, a new 3D US probe is introduced which can address the above mentioned limitations of 2D US for access procedures.

The investigators hypothesize that this superior three dimensional awareness can improve needle placement during central venous catheterization, increasing success rates and potentially decreasing complications.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiothoracic surgery with need for central venous catheter placement
* written informed consent

Exclusion Criteria:

* no informed consent
* other site for central line placement (eg subclavian vein)
* emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
first pass success | during procedure/surgery
  successful entry in internal jugular vein within one skin break and fluid motion

SECONDARY OUTCOMES:
imaging time | during procedure/surgery
  time from placing USprobe until start needling (in seconds)
needling time | during procedure/surgery
  time from puncturing skin until access in vein (in seconds)
number of skin punctures | during procedure/surgery
  total skin breaks needed before successful entry in vein
number of needle withdrawals | during procedure/surgery
  redirections of needle >5mm without needing new skin breaks
number of posterior wall punctures | during procedure/surgery
  puncture of posterior wall of jugular vein
operator satisfaction | procedure/surgery
  satisfaction of operator with visual feedback from US, rated on Likert Scale 1-5 with 1 no satisfaction at all and 5 totally satisfied
needle visibility | procedure/surgery
  visualization of needle during procedure on US screen, rating from good - adequate - poor

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scholten HJ, Meesters MI, Montenij LJ, Korsten EHM, Bouwman RA; 3DUI Study group. 3D biplane versus conventional 2D ultrasound imaging for internal jugular vein cannulation. Intensive Care Med. 2022 Feb;48(2):236-237. doi: 10.1007/s00134-021-06579-9. Epub 2021 Nov 22. No abstract available. PMID 34807306